CLINICAL TRIAL: NCT04456426
Title: Evaluation of the Characteristics of Patients With Suspected or Confirmed of COVID-19 in Villavicencio and Meta State, Colombia
Brief Title: Characteristics of Patients With COVID-19 in Meta State, Colombia
Status: Withdrawn | Type: Observational
Why Stopped: No access to the database of healthcare workers.
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Clínica Primavera (Unknown); Clínica Meta (Unknown); Cooperative University of Colombia (Other); Grupo de Investigación de Villavicencio (Unknown)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Critical Care Chief of Staff; professor of medicine, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2020_01COVID
Record Dates: First submitted 2020-05-29; First posted 2020-07-02 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: COVID; SARS-CoV 2; SARS Pneumonia; SARS (Disease); SARS (Severe Acute Respiratory Syndrome)
Keywords: COVID; SARS; Viral Pneumonia; SARS-CoV 2; Coronavirus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Disease; Pneumonia, Viral; Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with COVID-19: All populations of patients admitted with COVID-19 in healthcare institutions involved. No intervention but standard care designed by national guidelines will be provided.

SUMMARY:
This observational study aims to collect detailed clinical information on confirmed or suspected patients of COVID-19 treated in hospitals from Meta State, Colombia. The objectives are:

1. To establish the characteristics of patients and healthcare workers treated with COVID-19.
2. To assess previous predisposing morbidity.
3. To detail clinical factors associated with complications.
4. To profile clinical indicators for severity and outcomes.

DETAILED DESCRIPTION:
Hospital database and clinical charts in an electronic format of patients with suspected or confirmed COVID-19 will be reviewed to include in the study. Multiple centers from the eastern Colombian prairies caring for this population will participate to provide an understanding of the behavior of the epidemic and accurate clinical comprehension of the disease. Healthcare centers involved in providing an evaluation of patients infected with SARS-CoV-2 will be invited to participate.

The study will focus on the routine or new treatment strategies provided and a large population of patients analyzed would be desirable. It will allow identifying the most relevant factors associated with clinical outcomes, complications, and prognosis, with an appropriate statistical methodology for the analysis of observational nature.

Variables of individuals assisted will be recorded as well as the end results, such as baseline characteristics of individuals and disease, and main outcomes such as mortality, need for ICU attention, mechanical ventilation, and length of stay.

These results will be used to promote an improvement in the quality of care and individual and cluster decisions in the region.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to participant institutions with respiratory symptoms or diagnosed as compatible with COVID-19.

Exclusion Criteria:

* None.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with respiratory symptoms compatible with a disease which might eventually result to be COVID-19 or not.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Death within 30 days of hospital admission
ICU admission | 30 days
  Need for intensive care unit admission
Mechanical ventilation | 30 days
  Need for intubation and invasive mechanical ventilation

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Duration of stay in the intensive care unit
Hospital length of stay | 30 days
  Duration of stay in hospitalization
Days of mechanical ventilation | 30 days
  Duration of mechanical ventilation included with intubation or tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Study Director — Grupo de Investigación de Villavicencio

IPD SHARING:
Plan to Share IPD: Undecided
Mendeley Data

REFERENCES:
- [Result] Hui DSC, Zumla A. Severe Acute Respiratory Syndrome: Historical, Epidemiologic, and Clinical Features. Infect Dis Clin North Am. 2019 Dec;33(4):869-889. doi: 10.1016/j.idc.2019.07.001. PMID 31668196
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Result] McMichael TM, Currie DW, Clark S, Pogosjans S, Kay M, Schwartz NG, Lewis J, Baer A, Kawakami V, Lukoff MD, Ferro J, Brostrom-Smith C, Rea TD, Sayre MR, Riedo FX, Russell D, Hiatt B, Montgomery P, Rao AK, Chow EJ, Tobolowsky F, Hughes MJ, Bardossy AC, Oakley LP, Jacobs JR, Stone ND, Reddy SC, Jernigan JA, Honein MA, Clark TA, Duchin JS; Public Health-Seattle and King County, EvergreenHealth, and CDC COVID-19 Investigation Team. Epidemiology of Covid-19 in a Long-Term Care Facility in King County, Washington. N Engl J Med. 2020 May 21;382(21):2005-2011. doi: 10.1056/NEJMoa2005412. Epub 2020 Mar 27. PMID 32220208
- [Result] Page KR, Venkataramani M, Beyrer C, Polk S. Undocumented U.S. Immigrants and Covid-19. N Engl J Med. 2020 May 21;382(21):e62. doi: 10.1056/NEJMp2005953. Epub 2020 Mar 27. No abstract available. PMID 32220207
- [Result] Rosenbaum L. Facing Covid-19 in Italy - Ethics, Logistics, and Therapeutics on the Epidemic's Front Line. N Engl J Med. 2020 May 14;382(20):1873-1875. doi: 10.1056/NEJMp2005492. Epub 2020 Mar 18. No abstract available. PMID 32187459
- [Result] Porcheddu R, Serra C, Kelvin D, Kelvin N, Rubino S. Similarity in Case Fatality Rates (CFR) of COVID-19/SARS-COV-2 in Italy and China. J Infect Dev Ctries. 2020 Feb 29;14(2):125-128. doi: 10.3855/jidc.12600. PMID 32146445